CLINICAL TRIAL: NCT00895388
Title: Effects of Structured Rehabilitation Program on Quality of Life After Surgical Treatment for Rectal Cancer- a Randomized Controlled Clinical Trial
Brief Title: Effects of Structured Rehabilitation Program on Quality of Life in Rectal Cancer Patients- a Randomized Controlled Trial
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of North Norway (Other)
Collaborators: Helse Nord (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P REK NORD 105/2007
Record Dates: First submitted 2009-05-07; First posted 2009-05-08 (Estimated); Last update posted 2024-03-05 (Actual); Status verified 2011-11

CONDITIONS: Quality of Life; Sexual Function; Urinary Incontinence; Anal Incontinence
Keywords: Urinary function; Anal function
MeSH Terms: conditions — Urinary Incontinence; Encopresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Structured Rehabilitation program (Other)
  Interventions: Behavioral: Structured Rehabilitation program
- Controls (No Intervention)

INTERVENTIONS:
Behavioral: Structured Rehabilitation program — Questionnaire send by post at 3, 6, 12, 18 and 24 months after operation
  Arms: Structured Rehabilitation program

SUMMARY:
Quality of life after rectal surgery is reported to be impaired. Side effects of surgery and/or neoadjuvant treatment as functional disturbances like sexual dysfunction, urinary incontinence, anal incontinence or stoma problems are commonly experienced. The investigators hypotheses is that structured rehabilitation program addressing these problems will improve quality of life. A RCT are performed in order to document the effects of the rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Rectal cancer Surgically treated for rectal cancer Informed concent Included in national guidelines for surveillance of rectal cancer patients

Exclusion Criteria:

* Older than 75 years Mentally or physically not able to participate Non curative surgical treatment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-05; Primary Completion 2019-11 (Actual); Study Completion 2019-12-02 (Actual)

PRIMARY OUTCOMES:
Quality of Life (EORTC QLQ-C30, EORTC QLQ-CR38) | Baseline, 3, 6, 12,18 and 24 months postoperative.
Quality of LIfe (EQ 5D) | Baseline, 3,6,12, 18 and 24.

SECONDARY OUTCOMES:
St Marks incontinence | Baseline, 3, 12 and 24
ICIQ sexual function | baseline, 3,12 and 24
ICIQ Urinary function Short form | baseline,3, 12 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Rolv-Ole Lindsetmo, MD, Phd, Mph, Study Director — Dep of gastrointestinal surgery, University Hospital of North Norway
Locations (1):
- Dep. of gastrointestinal surgery, University Hospital of North Norway, Tromsø, Norway